CLINICAL TRIAL: NCT03367936
Title: 12 Months Weight Loss Study Using Feedback Messages Delivered Via Smartphone
Brief Title: Promoting Lifestyle Change Via Tailored mHealth Feedback to Improve Health
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lora Burke, Professor of Nursing and Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO17040453; 1R01HL131583-01A1 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2021-04

CONDITIONS: Overweight and Obesity
Keywords: mobile technology; feedback message; self-monitoring
MeSH Terms: conditions — Overweight; Obesity | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-monitoring group (Active Comparator): All subjects will use a smartphone to self-monitor diet and monitor physical activity (Fitbit Charge 2), and a Withings or Fitibit digital scale for weight. Following randomization, participants will be oriented to Self-monitoring and provided a tutorial with images shown on the laptop and devices as well as printed materials showing the screen shots. At baseline, each participant will have a one-on-one session with the project interventionist, which covers the core principles of behavioral weight loss. The participant also will be given personalized fat, calorie, and PA goals for weight loss and information about how to access the intervention materials from the Diabetes Prevention Program (DPP) online which is publicly available (https://www.diabetesprevention.pitt.edu/).
  Interventions: Behavioral: One-on-one Session; Behavioral: Self-monitoring
- Self-monitoring+Feedback group (Experimental): All subjects will be asked to do everything the self-monitoring group is asked to do. Subjects will receive up to 4 Feedback messages per day (messages will be delivered between the hours set by the participants on the participant's phone, e.g., 8 AM and 9:30 PM). Messages will be delivered automatically, remotely and in real-time. Messages will be tailored to each participant's progress based on standardized algorithms. The Feedback program will be explained to them and how this is responsive to information entered on the self-monitoring diaries.
  Interventions: Behavioral: One-on-one Session; Behavioral: Self-monitoring; Behavioral: Feedback

INTERVENTIONS:
Behavioral: One-on-one Session — Participants will receive a 45-minute one-on-one behavioral lifestyle program for a healthful lifestyle and weight loss.
Behavioral: Self-monitoring — Participants will receive an orientation on how to self-monitor using the smartphone and other devises
Behavioral: Feedback — Participants will receive up to 4 daily feedback messages based on progress in attaining target behavior. The feedback messages will be delivered on a variable ratio schedule and tailored to data in subjects' dietary recordings
  Arms: Self-monitoring+Feedback group

SUMMARY:
The overall purpose of this randomized clinical trial is to examine the effect and efficacy of the individualized, real-time, smartphone-based feedback of diet and physical activity self-monitoring on subsequent weight-control behaviors, weight loss outcomes and sustainability of patient engagement. Participants will be randomized to one of 2 groups: (1) Self-Monitoring -similar to what many people do on their own, subjects will self-monitor diet, physical activity using Fitbit and weight using a Bluetooth-enabled scale, and (2) Self-Monitoring +Feedback-participants will self-monitor as described for the Self-Monitoring group but also will receive tailored Feedback messages. The Self-Monitoring +Feedback participants will receive up to 4 daily discrete pop-up Feedback messages on the participant's smartphone delivered at random times during waking hours and tailored to content of recorded entries in the subjects' smartphone-based diaries and a weekly summary Feedback message about the participant's weight.

DETAILED DESCRIPTION:
This study includes the following activities:

1. Screening:

   Phase I: It will be conducted online. Respondents to recruitment solicitations will be provided an online Uniform Resource Locator (URL) with a hyperlink to a study flier that describes the essential elements of the study. It will also include a choice of URL or Quick Response (QR) code to access an online survey that will provide more details about the study. The research staff will also ask preliminary questions about eligibility (age, height and weight to calculate BMI), and consent to have the research team review the participant's answers.

   Phase II: It will be conducted online. After completing an online consent, the participants will provide personal information in the Sociodemographic and Lifestyle Questionnaire and health and medical conditions in the General Health History questionnaire as well as the Center for Epidemiologic Studies Depression Scale (CES-D) and the Eating Habits Checklist to screen for eating disorders.

   Run-in period: To minimize attrition and ensure that potential subjects are appropriate for the intervention, research staff will teach all eligible individuals how to download and complete a 5-day Self-Monitoring diary using the My Food Diary (Fitbit) Self-Monitoring program on the participant's phone or computer. After review of the diary, research staff will contact the potential participant to schedule the baseline assessment. Individuals need to record at least 700 kcal/day of food intake to be eligible for the study. Each user will have a username and password and also have the ability to manage the participant's own privacy settings.

   Baseline Assessment: Individuals who remain eligible will be invited to a screening appointment where the investigators measure the participant's height/weight for BMI, and explain the aims of the study and the 2 group conditions. If interested in participating, attendees will be asked to sign a consent form for the baseline data collection. At this visit, the participants will be asked to complete the Barriers to Healthy Eating scale; Weight Efficacy Lifestyle (WLE); Self-Efficacy and Eating Habits Survey; Self-Efficacy and Exercise Habits Survey; Self-Regulation of Eating Behavior Questionnaire; a one-page questionnaire (Quick WAVE140) that assesses current diet and PA habits, PROMIS Sleep Disturbance Short Form 8a; Effort-Reward Imbalance questionnaire; and ASA-24 Dietary Recall (two different days) . At the end of the baseline assessment, participants will be scheduled for a One-on-One session with a master's prepared registered dietician who will conduct an interview WAVE screener and provide counseling regarding lifestyle habits that support weight loss.
2. Randomization:

   At the One-on-One session, the research staff will use a computer software program on a laptop to determine to which group the individual will be randomized. (Prior to this time, the randomization scheme will be implemented via a computerized program (Visual Basic 6.0) using minimization method, which will be overseen by a statistician (Co-PI: S Sereika). Each of the 2 conditions (Self-Monitoring alone or Self-Monitoring plus Feedback) will be assigned a total of 265 subjects with randomization stratified by gender and race. After randomization, all participants will receive instructions on using the Fitbit Charge 2™ for physical activity and the Withings or Fitbit scale for self-weighing.
3. Intervention:

   The intervention will consist of the Self-Monitoring and Feedback program and remote guidance to a lifestyle program for weight loss. All participants will be subscribed to My Food Diary an online Self-Monitoring program that can be accessed via the participant's smartphone or any computer. The interventionists will have access to the diaries so the study staff can contact a participant if there is any safety concern about the reported eating behaviors. The study will provide all participants a wrist-worn FitBit Charge 2™ to self-monitor the participant's physical activity which synchs with the participant's phone or computer. The study will also provide all participants a Bluetooth-enabled scale (Withings or Fitbit) for self-monitoring the participant's weight. The Withings scale will transmit the weight values to the smartphone, Health Mate app and server, so the research team will know the weight status of participants. The Fitbit scale will transmit weights to the Fitbit server and then to the participant's phone so that study staff can monitor weight. The subject registers as the primary scale user and is subsequently recognized and distinguished from other household users. The scale displays the weight accurately to the 10th decimal. The data are converted to graphs for easy review. Batteries have a 6-12 month life. The scale measures weights between 5 and 180 kg. Participants will weigh themselves with the device daily; participants will be able to view the participant's weight data on the participant's smartphone. The Fitbit will provide data on daily steps and distance walked, which will be used to inform the selection of message that the investigators will provide participants in the Self-Monitoring plus Feedback group feedback messages related to physical activity. The data that will be transmitted between the Fitbit and Pitt servers will not contain any identifying personal information nor will Fitbit store any identifying information for the participants.

   Self-Monitoring group (Control Group): Individuals in this condition will not receive Feedback messages. All subjects will use a smartphone to self-monitor diet (My Food Diary), Fitbit Charge 2™ to monitor PA, and a Withings/Fitbit digital scale for weight. The Fitbit app is publically available. At the baseline visit following randomization, participants will be oriented to Self-Monitoring and the various Self-Monitoring devices and apps, and provided a tutorial with images shown on the laptop and devices as well as printed materials showing the screen shots. At this baseline session, each participant will have a one-on-one session with the project interventionist which covers the core principles of behavioral weight loss to ensure all understand basic recommendations for safe and effective weight loss. The participants also will be given personalized fat, calorie, and physical activity goals for weight loss and information about how to access the intervention materials from the Diabetes Prevention Program (DPP) online which is publicly available (https://www.diabetesprevention.pitt.edu/).

   Self-Monitoring+Feedback (Intervention Group)-This group will receive up to 4 Feedback messages per day (messages will be delivered between the hours set by the participants on the participant's phone, e.g., 8 AM and 9:30 PM). Messages will be delivered automatically, remotely and in real-time. it will be tailored to each participant's progress based on standardized algorithms. At the baseline visit following randomization, participants will be oriented to Self-Monitoring and the various Self-Monitoring devices and apps, and provided a tutorial with images shown on the laptop and devices as well as printed materials showing the screen shots. In addition, the Feedback program will be explained to them and how this is responsive to information entered on the Self-Monitoring diaries. Also, the participants will be given a brief handout on fat, calorie, physical activity and weight goals for weight loss and information about how to access the intervention materials from the Diabetes Prevention Program (DPP) online.

   The research team is able to review the Self-Monitoring data, and will check the data weekly. If any indication of rapid weight loss or periods of inactivity occur, research staff will contact the subject.
4. Measurements used in Study: At Phase I and II Screening: Medical and Weight History Form, Sociodemographic Form, Binge Eating Scale (Eating Habits Checklist), Center for Epidemiologic Studies Depression (CES-D); At baseline, 6 and 12 months: Weight (Withings or Fitbit scale, smartphone), blood pressure, waist circumference, Self-Regulation of Eating Behavior Questionnaire (SREBQ), Barriers to Healthy Eating (BHE), Weight Efficacy Lifestyle (WEL), Self- Efficacy and Eating Habits Survey, Self-Efficacy and Exercise Habits Survey, Quick WAVE Screener Questionnaire, PROMIS Sleep Disturbance, Effort-Reward Imbalance Questionnaire, diet (24-Hour Dietary Recall & smartphone), PA (The FitBit Charge 2™, smartphone), Intervention Satisfaction Questionnaire (at 12 months only).

ELIGIBILITY:
Inclusion Criteria:

1. Currently own and regularly use a smartphone
2. Age ≥18 years;
3. BMI > 27 and < 43; and
4. Successful completion of a 5-day electronic diary of food intake during a run-in period.

Exclusion Criteria:

1. Presence of an unstable condition requiring physician-supervised diet and exercise (e.g., recent myocardial infarction);
2. Physical limitations precluding ability to engage in moderate-intensity physical activity;
3. Pregnancy or intention to become pregnant during study;
4. Current treatment for a serious mental illness (e.g. schizophrenia);
5. Reported alcohol intake > 4 drinks/day;
6. Participation in a formal weight loss program, loss of ≥ 5% weight in past 6 month, or current use of weight loss medication;
7. History of bariatric surgery in <5 years,
8. Planned extended vacations, absences, or relocation during study;
9. A score >16 on the Center for Epidemiologic Studies Depression Scale (CES-D);
10. Score >32 on the Eating Habits Checklist, an eating disorder scale administered at baseline. For those who have an elevated BDI score (>22) or EHC (>32), we offer referral for counseling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6 and 12 months
  Changes in weight: measured as percent change in weight from baseline to 6 and 12 months

SECONDARY OUTCOMES:
Adherence to behavioral goals | 6 and 12 months
  Number of days participants met the dietary and physical activity goals
Adherence to self-weighing | 6 and 12 months
  Number of days participants self-weigh
Adherence to treatment protocol | 6 and 12 months
  Number of days participants self-monitor

OTHER OUTCOMES:
Retention | 6 and 12 months
  The percentage of participants who stay in the study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data.

REFERENCES:
- [Derived] Cheng J, Costacou T, Sereika SM, Conroy MB, Parmanto B, Rockette-Wagner B, Kriska AM, Klem ML, Burke LE. Effect of an mHealth weight loss intervention on Healthy Eating Index diet quality: the SMARTER randomised controlled trial. Br J Nutr. 2023 Dec 14;130(11):2013-2021. doi: 10.1017/S0007114523001137. Epub 2023 Jun 7. PMID 38713063
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Bizhanova Z, Sereika SM, Brooks MM, Rockette-Wagner B, Kariuki JK, Burke LE. Identifying Predictors of Adherence to the Physical Activity Goal: A Secondary Analysis of the SMARTER Weight Loss Trial. Med Sci Sports Exerc. 2023 May 1;55(5):856-864. doi: 10.1249/MSS.0000000000003114. Epub 2022 Dec 28. PMID 36574734
- [Derived] Burke LE, Sereika SM, Bizhanova Z, Parmanto B, Kariuki J, Cheng J, Beatrice B, Cedillo M, Pulantara IW, Wang Y, Loar I, Conroy MB. The Effect of Tailored, Daily, Smartphone Feedback to Lifestyle Self-Monitoring on Weight Loss at 12 Months: the SMARTER Randomized Clinical Trial. J Med Internet Res. 2022 Jul 5;24(7):e38243. doi: 10.2196/38243. PMID 35787516
- [Derived] Burke LE, Sereika SM, Parmanto B, Bizhanova Z, Kariuki JK, Cheng J, Beatrice B, Loar I, Pulantara IW, Wang Y, Cedillo M, Conroy MB. Effect of tailored, daily feedback with lifestyle self-monitoring on weight loss: The SMARTER randomized clinical trial. Obesity (Silver Spring). 2022 Jan;30(1):75-84. doi: 10.1002/oby.23321. Epub 2021 Dec 12. PMID 34898011